CLINICAL TRIAL: NCT03656172
Title: Investigating the Value of Reticulocyte Haemoglobin Content (RET-he) in the Management of Functional Martial Deficiency Anaemia in Patients With Solid Tumours
Brief Title: Interest of Reticulocyte Haemoglobin Content (RET-he) in Management of Functional Anemia for Patient With Solid Tumor
Acronym: RET-HE
Status: Completed | Type: Observational
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Other Study IDs: ICO-N-2017-01
Record Dates: First submitted 2018-08-28; First posted 2018-09-04 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Solid Tumor, Adult; Anemia Deficiency
Keywords: Anemia by functional martial deficiency; RET-He

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Haemoglobin measure: Anaemic adult Patients eligible to iron Treatment supported within the ICO for a solid tumor, untreated or treated by chemotherapy and/or radiotherapy and/or surgery, having benefited of a blood test (NFS, reticulocytes with RET-He , a martial blood test (iron, transferrin and Ferritin), a CRP, vitamins B12 and B9, a creatinine, a haptoglobin, a TSH) before and after iron treatment.
  Interventions: Biological: Haemoglobin measure

INTERVENTIONS:
Biological: Haemoglobin measure — Haemoglobin measure before and one month after standard iron treatment

SUMMARY:
Determine the value of the initial measurement of the hemoglobin content of reticulocytes (RET-He) for predicting the response to martial treatment for patients with a solid tumor with a functional martial deficiency as defined NCCN2016 (with or without inflammation). The aim is to refine the current definition of functional martial deficiency in order to best adapt the iron prescription in oncology by giving iron only if necessary, i.e. if the RET is low.

DETAILED DESCRIPTION:
Anemia is a common clinical situation in oncology. It contributes to the asthenia and thus to the decrease in the quality of life of the patient. In addition, it is considered an independent pejorative prognostic factor according to a literature review of 2001. An appropriate management of the latter is therefore paramount. To do this, it is necessary to successfully define its origins.

In 2014, RET-he was studied for the first time in the cancer patient. This analysis showed that there is a good negative predictive value of RET-he for a cut-off of 32 PG, i.e., that above this value the iron deficiency is unlikely. Iron deficiency anemia was defined by hemoglobin below 11 g/dl, serum iron less than 40 Μ g/dl, and TSAT less than 20%. However, this study had some limiting factors. First, patients were not separated according to cancer pathology: solid tumors versus malignant hemic. In addition, previous treatments, such as the administration of ASE, iron and/or globular pellets, have not been taken into account. The number of patients with anemia and iron deficiency was limited (n = 23). Despite these different biases, this study is the first to demonstrate the interest of this parameter in the management of anemia in the patient in oncology.

In total, the data are consistent with the potential interest of the hemoglobin content of reticulocytes in the diagnosis of martial deficiency. This is why the purpose of this project is to establish a RET-He study in anaemic patients with a solid tumor to determine if this endpoint could be included in a diagram of the management of anemia in oncology, particularly for To detect subpopulations (responder patient or not to iron IV) in patients with a functional martial deficiency.

Patients will be included as they are taken care of in the facility. A delay of about 3 months is necessary for the information to be complete and validated. The file will be taken out at regular intervals to inform the patient's follow-up.

The establishment of the therapy to correct anemia (administration of iron IV (associated or not to an ASE) is the responsibility of the referring physician or other prescriber doctor by delegation.

The different follow-up points for each patient will be the standard assessments made according to the NCCN recommendations:

* Assessment 1: between J21 (= 3 wk) and J35 (= 5 wk) after the introduction of a treatment (= J0) : the blood test must include at least one NFS and reticulocytes with RET-He (carried out in the ICO laboratory). This assessment will allow an intermediate evaluation of the effectiveness of the treatment by the doctor in order to envisage a possible implementation under ASE.
* Assessment 2: between J36 (= 6 wk) and J84 (= 12 wk) after the introduction of a treatment (= J0). The blood test must include at least one NFS (carried out in the ICO laboratory).

An exclusion from the protocol will be carried out in a second step if the patient receives a globular pellet transfusion between the initial blood test and the assessment 1. The results of the assessment 2 will not be taken into account if the patient has a transfusion between the assessment 1 and the assessment 2.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Metastatic solid tumor or not.
* Anemia by functional martial deficiency (as defined in the NCCN2016 recommendations):

  o Hb < 11 g/DL, TSAT < 20% and ferritinlike between 30 and 800 ng/ml
* Initial assessment of anemia carried out at the laboratory of Biopathology of the ICO

Exclusion Criteria:

* Patient with malignant hemopathy.
* Patient with chronic renal failure with an estimation of renal filtration rate according to the formula CKD-EPI < 60 ml/min/1.73 m².
* Patient with vitamin B12 deficiency, folate deficiency, hemolysis and/or hemoglobinopathy.
* Patient with active infection.
* Patient with bone marrow tumor. Confirmation by a osteo-medullary biopsy (BOM) or a myelogram is not necessary to exclude the patient.
* Patient who received ASE within two months prior to the initial blood test.
* Patient who received iron (oral or injectable) in the two months preceding the initial blood test.
* Patient who received a transfusion of globular pellets in the month preceding the initial blood test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with anaemia treated at the ICO for a solid tumour, not treated or treated with chemotherapy and/or radiotherapy and/or surgery, having benefited before the inclusion of a blood test including an NFS, reticulocytes with RET-He , a martial blood test (iron, transferrin and Ferritin), a CRP, vitamins B12 and B9, a creatinine, a haptoglobin, a TSH.
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2017-05-04 (Actual); Primary Completion 2020-05-11 (Actual); Study Completion 2020-05-11 (Actual)

PRIMARY OUTCOMES:
To assess the value of the initial measurement of reticulocyte haemoglobin content (RET-He) in predicting response to martial therapy | 1 month after inclusion
  Correlation between the value of RET-He on the initial blood test and the response to intravenous iron treatment at 1 month after start of this treatment.

SECONDARY OUTCOMES:
Assess the effectiveness of therapeutic management of martial deficiency anaemia with Intravenous iron (with or without an ESA: Erythropoiesis-Stimulating Agent) | 3 months after inclusion
  Calculation of the percentage of patients responding to the treatment with intravenous iron (associated or not to an ESA: erythropoiesis-stimulating agent) in case of functional martial deficiency.
Determine whether the percentage Hypo-He parameter, corresponding to the percentage of hypochromic red blood cells (MCHT less than 17 pg), is of interest in the diagnosis of the type of anaemia | 3 months after inclusion
  Calculation of the percentage of HypoHe threshold to obtain a good Positive Predictive Value (PPV) of martial deficiency and/or a good Negative Predictive Value (NPV) of no deficiency

CONTACTS AND LOCATIONS:
Overall Officials: Mathilde DUPE, MD, Principal Investigator — Institut de Cancérologie de l'Ouest
Locations (1):
- Institut de Cancérologie de l'Ouest, Saint-Herblain, France